CLINICAL TRIAL: NCT06506851
Title: Effects of Augmented Reality-based Rapid Blood Transfusion (Level-1®) Education on Nurse's Clinical Competency, Self-efficacy, and Educational Satisfaction: Randomised Controlled Trial
Brief Title: Effects of Augmented Reality-based Rapid Blood Transfusion (Level-1®)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023-06-084
Record Dates: First submitted 2024-06-12; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-06

CONDITIONS: Equipment and Supplies; Augmented Reality; Nurse's Role
Keywords: Augmented Reality; Education, Nursing; Blood Transfusion; Self-efficacy; Educational Satisfaction; Clinical Competency; Critical Care

STUDY DESIGN:
Intervention Model Description: Experimental Group (AR-based Training):
  Nurses receive AR-based training with Microsoft HoloLens 2®, immersing them in interactive simulations for hands-on learning.
  Control Group (Traditional Self-Learning):
  Nurses follow traditional guideline-based self-learning methods without augmented reality technology.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AR-based Training Group (Experimental): Practical nurses in this arm receive AR-based training using Microsoft HoloLens 2®. This training method incorporates augmented reality technology to provide immersive and interactive learning experiences, enhancing their proficiency in device utilization.
  Interventions: Other: AR-based Training with Microsoft HoloLens 2®
- Traditional Self-Learning Group (Sham Comparator): Practical nurses in this arm follow traditional guideline-based self-learning methods without augmented reality technology. They rely on conventional educational materials and guidelines for learning device utilization skills.
  Interventions: Other: Traditional Guideline-based Self-Learning

INTERVENTIONS:
Other: AR-based Training with Microsoft HoloLens 2® — Practical nurses in this group receive AR-based training using Microsoft HoloLens 2®. This training method incorporates augmented reality technology to provide immersive and interactive learning experiences, enhancing their proficiency in device utilization.
  Arms: AR-based Training Group
Other: Traditional Guideline-based Self-Learning — Practical nurses in this group follow traditional guideline-based self-learning methods without augmented reality technology. They rely on conventional educational materials and guidelines for learning device utilization skills.
  Arms: Traditional Self-Learning Group

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of AR-based training with traditional guideline-based self-learning in practical nurses without prior Level-1® experience. The main questions it aims to answer are:

Does AR-based training using Microsoft HoloLens 2® improve clinical performance compared to traditional guideline-based self-learning? Does AR-based training affect self-efficacy and educational satisfaction compared to traditional methods?

Participants will:

Receive AR-based training using Microsoft HoloLens 2® (experimental group) Follow traditional guideline-based self-learning (control group) Researchers will compare the AR-based training group to the traditional self-learning group to see if AR-based training leads to better clinical performance, higher self-efficacy, and greater educational satisfaction.

DETAILED DESCRIPTION:
In critical situations like hypovolemic shock, nurses must master skills for using devices like the Level-1® rapid infusion system. However, limited exposure poses challenges. Augmented reality (AR) offers a solution by providing realistic practice scenarios. While AR has shown effectiveness in cardiopulmonary resuscitation and intubation education, its application in Level-1® training remains underexplored.

This study was conducted at the Samsung Medical Center in Seoul, Korea, and involved 42 practical nurses without prior Level-1® experience. Participants were randomly assigned to one of two groups: the experimental group, which received AR-based training using Microsoft HoloLens 2®, and the control group, which followed traditional guideline-based self-learning.

The study aimed to investigate the impact of AR-based Level-1® education on nurses' clinical performance, self-efficacy, and educational satisfaction. Clinical performance, self-efficacy, and educational satisfaction were assessed through structured measurements.

Results data and conclusions drawn from the data are excluded from this section and will be reported separately in the Results Section of the record.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate voluntarily and understanding of the study's purpose.
* No prior experience with the Level-1® rapid infusion system.

Exclusion Criteria:

* Failure to meet the inclusion criteria.
* Prior experience with the Level-1® rapid infusion system.
* Inability to comprehend the study's purpose or express voluntary participation.
* Inability to attend required training and evaluations.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2023-09-05 (Actual)

PRIMARY OUTCOMES:
Clinical Competency | before training, immediately after training
  This measurement assesses nurses' clinical competency in rapid infusion procedures. It includes evaluation of learning time, performance time, accuracy, and assistance requests.

SECONDARY OUTCOMES:
Self-efficacy | efore training, immediately after training
  This assessment measures nurses' self-efficacy in rapid infusion procedures using a modified self-efficacy scale. It evaluates confidence levels in performing tasks related to rapid infusion.

OTHER OUTCOMES:
Educational Satisfaction Evaluation | Educational satisfaction will be assessed immediately after the completion of the training program.
  This evaluation assesses nurses' satisfaction with the educational program. It includes measures of confidence, relevance, and willingness to recommend the training to others using a structured questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: meonghi son, MD, Study Chair — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea